CLINICAL TRIAL: NCT05914116
Title: A Phase 1/2a, Multicenter, Open-Label, First in Human Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of DB-1311 in Subjects With Advanced/Metastatic Solid Tumors
Brief Title: A Phase 1/2a Study of DB-1311/BNT324 in Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: DualityBio Inc. (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DB-1311-O-1001
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumors
Keywords: B7-H3; SCLC (small cell lung cancer); NSCLC (non-small cell lung cancer); ESCC (esophageal squamous cell carcinoma); CRPC (castration-resistant prostate cancer); Melanoma; HCC (Hepatocellular Carcinoma); HNSCC (Head and neck squamous cell carcinomas); CC (Cervical Cancer); PROC (platinum-resistant ovarian cancer); PC (prostate cancer); CSPC (castration-sensitive prostate cancer)
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Esophageal Squamous Cell Carcinoma; Melanoma; Carcinoma, Hepatocellular; Squamous Cell Carcinoma of Head and Neck; Uterine Cervical Neoplasms; Prostatic Neoplasms | interventions — Lopinavir; Ritonavir; Itraconazole; enzalutamide; abiraterone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (23):
- DB-1311/BNT324 Dose Level 1 (Experimental): Enrolled Subjects will receive a single-dose of DB-1311/BNT324 at Dose Level 1 on Day 1 of each cycle Q3W (every 3 weeks)
  Interventions: Drug: DB-1311
- DB-1311/BNT324 Dose Level 2 (Experimental): Enrolled Subjects will receive a single-dose of DB-1311/BNT324 at Dose Level 2 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1311
- DB-1311/BNT324 Dose Level 3 (Experimental): Enrolled Subjects will receive a single-dose of DB-1311/BNT324 at Dose Level 3 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1311
- DB-1311/BNT324 Dose Level 4 (Experimental): Enrolled Subjects will receive a single-dose of DB-1311/BNT324 at Dose Level 4 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1311
- DB-1311/BNT324 Dose Level 5 (Experimental): Enrolled Subjects will receive a single-dose of DB-1311/BNT324 at Dose Level 5 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1311
- DB-1311/BNT324 Dose Expansion 1 (Experimental): Subjects with advanced/unresectable, or metastatic SCLC who have progressed on or after standard systemic treatments, a 21-day treatment cycle (i.e., once every 3 weeks) via intravenous infusion will be used for DB-1311/BNT324 randomized at dose level 1 or 2.
  Interventions: Drug: DB-1311
- DB-1311/BNT324 Dose Expansion 2 (Experimental): Subjects with advanced/unresectable, or metastatic NSCLC who have progressed on or after standard systemic treatments, a 21-day treatment cycle (i.e., once every 3 weeks) via intravenous infusion will be used for DB-1311/BNT324 randomized at dose level 1 or 2.
  Interventions: Drug: DB-1311
- DB-1311/BNT324 Dose Expansion 3 (Experimental): Subjects with advanced/unresectable, or metastatic ESCC who have progressed on or after standard systemic treatments, a 21-day treatment cycle (i.e., once every 3 weeks) via intravenous infusion will be used for DB-1311/BNT324.
  Interventions: Drug: DB-1311
- DB-1311/BNT324 Dose Expansion 4 (Experimental): Subjects with advanced/unresectable, or metastatic CRPC who have progressed on or after standard systemic treatments, a 21-day treatment cycle (i.e., once every 3 weeks) via intravenous infusion will be used for DB-1311/BNT324 randomized at dose level 1 or 2.
  Interventions: Drug: DB-1311
- DB-1311/BNT324 Dose Expansion 5 (Experimental): Subjects with advanced/unresectable, or metastatic melanoma who have progressed on or after standard systemic treatments, a 21-day treatment cycle (i.e., once every 3 weeks) via intravenous infusion will be used for DB-1311/BNT324.
  Interventions: Drug: DB-1311
- DB-1311/BNT324 Dose Expansion 6 (Experimental): Subjects with advanced/unresectable, or metastatic HCC who have progressed on or after standard systemic treatments, a 21-day treatment cycle (i.e., once every 3 weeks) via intravenous infusion will be used for DB-1311/BNT324.
  Interventions: Drug: DB-1311
- DB-1311/BNT324 Dose Expansion 7 (Experimental): Subjects with advanced/unresectable, or metastatic cervical cancer who have progressed on or after standard systemic treatments, a 21-day treatment cycle (i.e., once every 3 weeks) via intravenous infusion will be used for DB-1311/BNT324.
  Interventions: Drug: DB-1311
- DB-1311/BNT324 Dose Expansion 8 (Experimental): Subjects with other advanced or metastatic solid tumors who have progressed on or after standard systemic treatments, a 21-day treatment cycle (i.e., once every 3 weeks) via intravenous infusion will be used for DB-1311/BNT324.
  Interventions: Drug: DB-1311
- DB-1311/BNT324 Dose Expansion 9 (Experimental): Subjects with advanced/unresectable, or metastatic HNSCC (not including nasopharyngeal carcinoma [NPC]) who have progressed on or after standard systemic treatments, a 21-day treatment cycle (i.e., once every 3 weeks) via intravenous infusion will be used for DB-1311/BNT324.
  Interventions: Drug: DB-1311
- DB-1311/BNT324 Dose Expansion 10 (Experimental): Subjects with advanced or metastatic rare tumor types who have progressed on or after standard systemic treatments, a 21-day treatment cycle (i.e., once every 3 weeks) via intravenous infusion will be used for DB-1311/BNT324.
  Interventions: Drug: DB-1311
- DB-1311/BNT324 Dose Expansion 11 (Experimental): Subjects with metastatic CRPC who have progressed on or after standard systemic treatments including no more than 2 lines of systemic chemotherapy, novel hormone therapy and lutetium-177 radioligand therapy, a 21-day treatment cycle (i.e., once every 3 weeks) via intravenous infusion will be used for DB-1311/BNT324.
  Interventions: Drug: DB-1311
- DB-1311/BNT324 Dose Expansion 12 (Experimental): Taxane-naive subjects with metastatic CRPC who have progressed on or after novel hormone therapy, a 21-day treatment cycle (i.e., once every 3 weeks) via intravenous infusion will be used for DB-1311/BNT324.
  Interventions: Drug: DB-1311
- DB-1311/BNT324 Dose Expansion 13 (Experimental): Subjects with advanced/unresectable, or metastatic HNSCC (not including NPC) who have progressed on or after standard systemic treatments, a 21-day treatment cycle (i.e., once every 3 weeks) via intravenous infusion will be used for DB-1311/BNT324.
  Interventions: Drug: DB-1311
- DB-1311/BNT324 Dose Expansion 14 (Experimental): Subjects with epithelial OC who have had 1-3 prior lines of systemic treatment and are platinum-resistant, a 21-day treatment cycle (i.e., once every 3 weeks) via intravenous infusion will be used for DB-1311/BNT324 randomized at dose level 1 or 2.
  Interventions: Drug: DB-1311
- DB-1311/BNT324 Dose Expansion 15 (Experimental): Subjects with Subjects with advanced/unresectable, or metastatic melanoma, ESCC, PROC and CC who have progressed on or after standard systemic treatments, a 21-day treatment cycle (i.e., once every 3 weeks) via IV will be used for DB-1311/BNT324.
  Lopinavir and ritonavir/ Itraconazole will be administered orally twice a day/ once a day.
  Interventions: Drug: DB-1311; Drug: Lopinavir and Ritonavir Tablets; Drug: itraconazole
- DB-1311/BNT324 Dose Expansion 16 (Experimental): Taxane-naive subjects with metastatic CRPC who have progressed on or after NHT, a 21-day treatment cycle (i.e., once every 3 weeks) via intravenous infusion will be used for DB-1311/BNT324, combined with enzalutamide 160mg QD orally.
  Interventions: Drug: DB-1311; Drug: Enzalutamide
- DB-1311/BNT324 Dose Expansion 17 (Experimental): Taxane-naive subjects with metastatic CRPC who have progressed on or after NHT, a 21-day treatment cycle (i.e., once every 3 weeks) via intravenous infusion will be used for DB-1311/BNT324, combined with abiraterone 1000mg QD orally.
  Interventions: Drug: DB-1311; Drug: Abiraterone
- DB-1311/BNT324 Dose Expansion 18 (Experimental): CSPC subjects with suboptimal PSA response to ADT/NHT, a 21-day treatment cycle (i.e., once every 3 weeks) via intravenous infusion will be used for DB-1311/BNT324, combined with enzalutamide 160mg or abiraterone 1000mg QD orally.
  Interventions: Drug: DB-1311; Drug: Enzalutamide; Drug: Abiraterone

INTERVENTIONS:
Drug: DB-1311 — Administered I.V.(intravenous infusion)
Drug: Lopinavir and Ritonavir Tablets — Lopinavir and Ritonavir Tablets
  Arms: DB-1311/BNT324 Dose Expansion 15
Drug: itraconazole — itraconazole
  Arms: DB-1311/BNT324 Dose Expansion 15
Drug: Enzalutamide — oral administration
  Arms: DB-1311/BNT324 Dose Expansion 16; DB-1311/BNT324 Dose Expansion 18
Drug: Abiraterone — oral administration
  Arms: DB-1311/BNT324 Dose Expansion 17; DB-1311/BNT324 Dose Expansion 18

SUMMARY:
This is a dose-escalation and dose-expansion Phase 1/2a trial to evaluate the safety and tolerability of DB-1311/BNT324 in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, open-label, multiple-dose, FIH Phase 1/2a study. Phase 1 adopts an accelerated titration at first dose level followed with classic "3+3" design to identify the MTD (maximum tolerated dose) and/or RP2D(Recommended Phase 2 Dose). Phase 2a is a dose expansion phase to confirm the safety, tolerability and explore efficacy in selected malignant solid tumors treated with DB-1311/BNT324 as monotherapy or in combination with novel hormone therapy (NHT) in prostate cancer (PC). And the drug-drug-interaction (DDI) sub-study to evaluate the effect of lopinavir/ritonavir and itraconazole on the PK of DB-1311 and its payload.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults (defined as ≥ 18 years of age or acceptable age according to local regulations at the time of voluntarily signing of informed consent).
2. Histologically or cytologically confirmed unresectable advanced/metastatic solid tumor that has relapsed or progressed on or after standard systemic treatments, or is intolerable with standard treatment; or for which no standard treatment is available.
3. At least one measurable lesion as assessed by the investigator according to response evaluation criteria in solid tumors (RECIST) version 1.1 criteria (measurable disease as defined by RANO 2.0 criteria for GBM subjects). Castrate-resistant prostate cancer (CRPC) subjects with bone only disease may be eligible on a case-by- case basis after discussion with the Medical Monitor.
4. Has a life expectancy of ≥ 3 months.
5. Has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1.
6. Has LVEF ≥ 50% by either echocardiography (ECHO) or multiple-gated acquisition (MUGA) within 28 days before enrollment.
7. Has adequate organ function within 7 days prior to Day 1 of Cycle 1
8. Has adequate treatment washout period prior to Day 1 of Cycle 1
9. Is willing to provide pre-existing resected tumor samples or undergo fresh tumor biopsy for the measurement of B7-H3 level and other biomarkers if no contraindication.

   Note: there is no minimum B7-H3 expression level mandatory for entry into the study.
10. Is capable of comprehending study procedures and risks outlined in the informed consent and able to provide written consent and agree to comply with the requirements of the study and the schedule of assessments.
11. Male and female subjects of reproductive/childbearing potential must agree to use adequate contraceptive methods (e.g., double barrier or intrauterine contraceptive) during the study and for at least 4 months and 7 months after the last dose of study drug, respectively.
12. Male subjects must not freeze or donate sperm starting at screening and throughout the study period, and at least 4 months after the final study drug administration.
13. Female subjects must not donate, or retrieve for their own use, ova from the time of screening and throughout the study treatment period, and for at least 7 months after the final study drug administration.
14. SCLC subjects (Phase 2a Cohort 1 ONLY):

    * Pathologically documented locally advanced, or metastatic SCLC not amenable to curative surgery or radiation.
    * Prior therapy with at least one platinum-based line as systemic therapy for extensive stage disease with at least two cycles of therapy (except in the case of early objective PD).
    * Prior treatment regimens with irinotecan, topotecan or any other TOP I inhibitor including investigational TOP I inhibitors are not allowed.
15. NSCLC subjects (Phase 2a Cohort 2 ONLY):

    * Pathologically documented locally advanced, or metastatic NSCLC and is not amenable to curative surgery or radiation.
    * Has received prior treatment with platinum-based chemotherapy regimen and/or anti-PD-1/PD-L1 antibody-based regimen in the advanced/unresectable, or metastatic setting unless unable or unwilling. Subjects with NSCLC known to harbor a genomic alteration(s) other than EGFR mutation(s) (e.g., ALK rearrangement, ROS1 rearrangement, KRAS G12C mutation, BRAF V600E mutation, NTRK1/2/3 Gene fusion, MET Exon 14 skipping, RET rearrangement etc.) for which treatment is available must have also received prior treatment with at least 1 genotype-directed therapy.
16. ESCC subjects (Phase 2a Cohort 3 ONLY):

    * Pathologically documented locally advanced, or metastatic ESCC and is not amenable to curative surgery or radiation.
    * Having received at least one prior therapy for unresectable disease. Patients with recurrence within 6 months of completion of neoadjuvant or adjuvant therapy will be considered as having received one prior therapy for unresectable disease.
17. CRPC subjects (Phase 2a Cohort 4 ONLY):

    • Pathologically documented metastatic adenocarcinoma of the prostate cancer.
    * Progressive metastatic CRPC as defined: 1) castrate levels of serum testosterone < 50 ng/dL AND 2) progressive disease as defined by PCWG3 criteria.
    * Having received prior docetaxel (before or after an AR-targeted therapy). Docetaxel rechallenge was allowed.
    * Having received prior novel hormone therapy.
18. Melanoma subjects (Phase 2a Cohort 5 ONLY) • Histologically or cytologically confirmed diagnosis of unresectable Stage III or metastatic melanoma not amenable to local therapy, must have had either:

    > Previously treated with a PD-1 or PD-L1 inhibitor.

    > If subjects with BRAF gene mutant melanoma, must have had a prior treatment regimen that included vemurafenib, dabrafenib, or another BRAF gene and/or mitogen-activated protein kinase (MEK) protein inhibitor.
19. HCC subjects (Phase 2a Cohort 6 ONLY)

    * Histological/cytological confirmed diagnosis of HCC or clinically confirmed diagnosis of HCC as per American Association for the Study of Liver Diseases (AASLD) criteria (fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC are not eligible), and:
    * Has received 1 or 2 prior systemic therapy regimens for recurrent or metastatic disease;
    * Has experienced disease progression during or after treatment with an anti-PD-1/L1 agent administered either as monotherapy or in combination.

    Note: Subjects basically should receive prior standard therapy.

    • However, if the investigator judges the therapy is not appropriate for the subject, the prior standard therapy is not necessarily mandated for the eligibility.

    • Has a Child-Pugh class A liver score within 7 days of first dose of study drug.
20. Cervical cancer subjects (Phase 2a Cohort 7 ONLY) • Has recurrent or metastatic cervical cancer with squamous cell, adenocarcinoma, or adenosquamous histology, and:

    • Has experienced disease progression during or after treatment with a standard of care systemic chemotherapy doublet, or platinum-based therapy (if eligible), defined as either: d. paclitaxel + cisplatin + bevacizumab + anti-PD-(L)1 agent, or e. paclitaxel + carboplatin + bevacizumab + anti-PD-(L)1 agent, or f. paclitaxel + topotecan + bevacizumab + anti-PD-(L)1 agent Note: In cases where bevacizumab and/or anti-PD-(L)1 agent is not a standard of care therapy or the subject was ineligible for such treatment according to local standards, prior treatment with bevacizumab and/or anti-PD-(L)1 agent is not required.

    • Has received 1 or 2 prior systemic therapy regimens for recurrent or metastatic cervical cancer. Chemotherapy administered in the adjuvant or neoadjuvant setting, or in combination with radiation therapy, should not be counted as a systemic therapy regimen. Single agent therapy with an anti-PD(L)1 agent for recurrent or metastatic cervical cancer should be counted.
21. Subjects with other solid tumors (Phase 2a Cohort 8 ONLY) • Histologically or cytologically confirmed solid tumors. • Progressed or relapsed after at least one prior standard therapeutic regimen (Patients who have not received all approved or standard treatments for their cancer must be informed that these alternatives to receiving DB-1311/BNT324 are available prior to consenting to participate in this trial).
22. HNSCC subjects (Phase 2a Cohort 9 and Cohort 13)

    • Histologically or cytologically confirmed refractory/metastatic (R/M) HNSCC (not including NPC) that is considered incurable by local therapies.

    • Progressed on or after prior standard therapeutic regimen.
23. Subjects with rare tumors (Phase 2a Cohort 10 ONLY) Histologically or cytologically confirmed rare tumor types. Progressed or relapsed after at least one prior standard therapeutic regimen (Patients who have not received all approved or standard treatments for their cancer must be informed that these alternatives to receiving DB-1311/BNT324 are available prior to consenting to participate in this trial).
24. Post lutetium-177 CRPC subjects (Phase 2a Cohort 11 ONLY):

    Pathologically documented metastatic adenocarcinoma of the prostate cancer. Progressive metastatic CRPC as defined: 1) castrate levels of serum testosterone < 50 ng/dL AND 2) progressive disease as defined by PCWG3 criteria.
25. Taxane-naive CRPC subjects (Phase 2a Cohort 12, 16, 17 ONLY)

    * Pathologically documented metastatic adenocarcinoma of the prostate cancer. Progressive metastatic CRPC as defined: 1) castrate levels of serum testosterone < 50 ng/dL AND 2) progressive disease as defined by PCWG3 criteria.

      26, PROC subjects (Phase 2a Cohort 14 ONLY)
    * Subjects must have a confirmed diagnosis of OC, primary peritoneal cancer, or fallopian tube cancer, all of which with high-grade serous or endometrioid histology..
    * Subjects must have platinum-resistant disease:
    * Received at least 1 but ≤ 3 lines of prior systemic anticancer therapy and have radiographic progressed on or after their most recent line of therapy.

27. CSPC with suboptimal PSA response (Phase 2a Cohort 18 ONLY)

* Pathologically documented adenocarcinoma of the prostate cancer.
* Having advanced/unresectable, or metastatic disease and confirmed by imaging (e.g., CT and/or bone scan).
* Having received ADT and enzalutamide or abiraterone for ≥4 months, with suboptimal PSA response.

  28. Additional inclusion criteria for DDI cohort: has a study treatment expectancy of >= 2.5 months. Able to withhold CYP3A/P-gp/OATP1B inhibitors or substrates or CYP3A inducers as concomitant treatments for certain period.

Exclusion Criteria:

Unless otherwise specified, the exclusion criteria are common to both Phase 1 and Phase 2a. Subjects who meet any of the following criteria will be excluded from the study:

1. Prior treatment with B7-H3 targeted therapy.
2. Prior treatment with antibody drug conjugate with topoisomerase inhibitor (e.g., trastuzumab deruxtecan).
3. Has a medical history of symptomatic congestive heart failure (CHF) (New York Heart Association [NYHA] classes II-IV) or serious cardiac arrhythmia requiring treatment.
4. Has a medical history of myocardial infarction or unstable angina within 6 months before enrollment.
5. Has an average of Fredericia's formula-QT corrected interval (QTcF) prolongation to > 470 millisecond (ms) in males and females based on a 12-lead electrocardiogram (ECG) in triplicate.
6. Use of concomitant medications known to prolong the QT interval. If the use is deemed necessary, they should be administered with caution and closely monitoring the QT interval, after discussed with the Sponsor.
7. Has a medical history of interstitial lung diseases (e.g., non-infectious interstitial pneumonia, pneumonitis, pulmonary fibrosis, and severe radiation pneumonitis) or current interstitial lung diseases or who are suspected to have these diseases by imaging at screening.
8. Has a history of underlying pulmonary disorder including, but not limited to, pulmonary emboli within 3 months of the start of study treatment, severe asthma, severe COPD, restrictive lung disease, and other clinically significant pulmonary compromise or requirement for supplemental oxygen.
9. Clinically significant gastrointestinal disorder including, but not limited to, history of gastrointestinal fistulation that need long-term intravenous nutrition; gastrointestinal dysfunction that need long-term enteral nutrition through the tube feeding; gastrointestinal obstruction/perforation that not recovered within 6 months prior to the enrollment.
10. Untreated or incompletely treated esophageal and/or gastric varices with bleeding or high risk of bleeding; A prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study treatment (Only applicable to HCC patients).
11. Metastatic disease that involves major airways or blood vessels (e.g., patients with vascular invasion of the major portal vein and inferior vena cava).
12. Clinically uncontrolled pleural effusion, ascites or pericardial effusion requiring drainage, peritoneal shunt or cell-free concentrated ascites reinfusion therapy within 2 weeks prior to the enrollment.
13. Any autoimmune, connective tissue or inflammatory disorders (e.g., rheumatoid arthritis, Sjögren's, sarcoidosis) where there is documented, or a suspicion of pulmonary involvement at the time of screening.
14. Has an uncontrolled infection requiring intravenous injection of antibiotics, antivirals, or antifungals.
15. Know human immunodeficiency virus (HIV) infection.
16. Subjects have active viral (any etiology) hepatitis are excluded. However, subjects with serologic evidence of chronic hepatitis B virus (HBV) infection (defined by a positive hepatitis B surface antigen [HBsAg] test or a positive hepatitis B core antibody test) who have a viral load below the limit quantification (e.g., HBV DNA titer < 1000 cps/mL or 200 IU/mL) and are willing to and maintain antiviral treatment if required, are eligible. However, subjects with a history of hepatitis C virus (HCV) infection who have completed curative antiviral treatment and have a viral load below the limit of quantification are eligible for study entry.
17. Is a lactating mother (women who are willing to temporarily interrupt breastfeeding will also be excluded), or pregnant as confirmed by pregnancy tests performed within 7 days prior to enrollment.
18. Has spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms. Subjects with clinically inactive brain metastases may be included in the study. Subjects with treated brain metastases that are no longer symptomatic and who require no treatment with corticosteroids or anticonvulsants may be included in the study if they have recovered from the acute toxic effect of radiotherapy. A minimum of 2 weeks must have elapsed between the end of whole brain radiotherapy and study randomization.
19. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to NCI-CTCAE version 5.0, grade ≤ 1 or baseline. Subjects with chronic Grade 2 toxicities (e.g., Grade 2 neuropathy) may be eligible based on the discussion and agreement between Investigator and Sponsor.
20. Has multiple primary malignancies within 3 years before enrollment, except adequately resected non-melanoma skin cancer (e.g., resected basal or squamous cell skin cancer), curatively treated in-situ disease (e.g., carcinoma in situ of the cervix or breast), other solid tumors curatively treated (e.g., superficial bladder cancer), or contralateral breast cancer.
21. Has substance abuse or any other medical conditions that would increase the safety risk to the subject or interfere with participation or evaluation of the clinical study in the opinion of the investigator.
22. Has known hypersensitivity to either the drug substances or inactive ingredients in the drug product.
23. Patients with other reasons that, in the opinion of the Investigator, make them unsuitable to participate in this study.
24. Additional exclusion criteria for DDI cohort: Has a contraindication for receiving lopinavir, ritonavir or itraconazole according to the prescribing information is not able to take lopinavir, ritonavir or itraconazole by oral intake.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 862 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Percentage of Participants with Dose-Limiting Toxicities (DLTs) as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Percentage of participants in Part 1 with DLTs | up to 21 days after Cycle 1 Day 1
  Percentage of participants in Part 1 with DLTs
Phase 1& Phase 2a: Percentage of Participants with Treatment Emergent Adverse Events (TEAEs) as assessed by CTCAE v5.0. | Up to follow-up period, approximately 1 year post-treatment
  Percentage of participants with TEAEs graded according to National Cancer Institute (NCI) CTCAE v5.0
Phase 1& Phase 2a: Percentage of Participants with Serious Adverse Events (SAEs) as assessed by CTCAE v5.0. | Up to follow-up period, approximately 1 year post-treatment
  Percentage of Participants with SAEs graded according to NCI CTCAE v5.0
Phase 1 & Phase 2a: vital sign measurements | Up to follow-up period, approximately 1 year post-treatment
Phase 1& Phase 2a: clinical safety laboratory parameters | Up to follow-up period, approximately 1 year post-treatment
Phase 1& Phase 2a: Electrocardiogram (ECG) parameters | Up to follow-up period, approximately 1 year post-treatment
Phase 1& Phase 2a: Eastern Cooperative Oncology Group (ECOG) performance status (PS) | Up to follow-up period, approximately 1 year post-treatment
Phase 1& Phase 2a: left ventricular ejection fraction (LEVF) | Up to follow-up period, approximately 1 year post-treatment
Phase 1: Maximum Tolerated Dose (MTD) of DB-1311/BNT324 | Up to the completion of Part 1 (assessed up to 12 months)
  MTD on the data collected during Part 1
Phase 1: Recommended Phase 2 Dose (RP2D) of DB-1311/BNT324 | Up to the completion of Part 1 (assessed up to 12 months)
  RP2D of DB-1311/BNT324 based on the data collected during Part 1
Phase 2a: Objective Response Rate (ORR) as determined by investigator | Up to follow-up period, approximately 1 year post-treatment
  Objective Response Rate (ORR) as determined by investigator per RECIST 1.1 in non-PC/non-GBM participants per RECIST v1.1 for soft tissue and Prostate Cancer Working Group 3 (PCWG3) criteria for bone metastases in PC participants, and ORR per neuro-oncology 2.0 (RANO 2.0) criteria in GBM participants.

SECONDARY OUTCOMES:
Phase 1: Objective response rate (ORR) | Up to follow-up period, approximately 1 year post-treatment
  ORR will be determined by investigator per RECIST v1.1 in non-CRPC participants, and per RECIST v1.1 for soft tissue and PCWG3 criteria for bone metastases in CRPC participants
Phase 1 & Phase 2a: duration of response (DoR) | Up to follow-up period, approximately 1 year post-treatment
  DoR will be determined by investigator per RECIST v1.1 in non-PC/non-GBM participants, per RECIST v1.1 for soft tissue and PCWG3 criteria for bone metastases in PC participants, and per RANO 2.0 criteria in GBM participants
Phase 1 & Phase 2a: disease-control rate (DCR) | Up to follow-up period, approximately 1 year post-treatment
  DCR will be determined by investigator per RECIST v1.1 in non-PC/non-GBM participants, per RECIST v1.1 for soft tissue and PCWG3 criteria for bone metastases in PC participants, and per RANO 2.0 criteria in GBM participants
Phase 1 & Phase 2a: Time to Response (TTR) | Up to follow-up period, approximately 1 year post-treatment
  TTR will be determined by investigator per RECIST v1.1 in non-PC/non-GBM participants, per RECIST v1.1 for soft tissue and PCWG3 criteria for bone metastases in PC participants, and per RANO 2.0 criteria in GBM participants
Phase 1 & Phase 2a: Progression Free Survival (PFS) | Up to follow-up period, approximately 1 year post-treatment
  PFS will be determined by investigator per RECIST v1.1 in non-PC/non-GBM participants, and per RANO 2.0 criteria in GBM participants
Phase 1 & Phase 2a: Radiographic Progression Free Survival (rPFS) | Up to follow-up period, approximately 1 year post-treatment
  rPFS will be determined by investigator per RECIST v1.1 for soft tissue and PCWG3 criteria for bone metastases in PC participants
Phase 1 & Phase 2a: Overall Survival (OS) | From date of first dose until the date of death or lost to follow up, approximately 1 year post-treatment
  OS is defined as the time from date of first dose to the date of death.
Phase 2a: Prostate-specific antigen (PSA) | From date of first dose until the date of first PSA progression, approximately 1 year post-treatment
  Time to PSA progression, PSA50 response rate and PSA90 response rate, duration of PSA response in PC participants and the rate of PSA conversion to <0.2 in CSPC.
Phase 2a: CA-125 response rate | Up to follow-up period, approximately 1 year post-treatment
  CA-125 response assessed per GCIG criteria for ovarian cancer subjects
Phase 1 & Phase 2a: Pharmacokinetic-AUC | within 8 cycles (each cycle is 21 days)
  Area under the concentration-time curve from time 0 to infinity of DB-1311/BNT324 ADC, total anti-B7-H3 antibody, and unconjugated P1021
Phase 1 & Phase 2a: Pharmacokinetic-Cmax | within 8 cycles (each cycle is 21 days)
  Maximum observed plasma concentration (Cmax) of DB-1311/BNT324 ADC, total anti-B7-H3 antibody, and unconjugated P1021
Phase 1 & Phase 2a: Pharmacokinetic-Tmax | within 8 cycles (each cycle is 21 days)
  Time to Cmax of DB-1311/BNT324 ADC, total anti-B7-H3 antibody, and unconjugated P1021
Phase 1 & Phase 2a: Pharmacokinetic-Cthrough | within 8 cycles (each cycle is 21 days)
  Trough concentration
Phase 1 & 2a: Anti-drug antibody (ADA) prevalence | Up to follow-up period, approximately 1 year post-treatment
  Percentage of participants who are ADA positive at any point
Phase 1 & 2a: ADA incidence | Up to follow-up period, approximately 1 year post-treatment
  Percentage of participants having treatment-emergent ADA

CONTACTS AND LOCATIONS:
Overall Officials: Lily Hu, Study Director — DualityBio Inc.
Locations (107):
- United States (28):
  - Research Site 111, Tucson, Arizona
  - Research Site 125, Los Angeles, California
  - Research Site 133, Los Angeles, California
  - Research Site 103, Los Angeles, California
  - Research Site 128, Santa Monica, California
  - Research Site 118, Celebration, Florida
  - Research Site 127, Margate, Florida
  - Research Site 137, Orlando, Florida
  - Research Site 101, Plantation, Florida
  - Research Site 109, Tamarac, Florida
  - Research Site 114, Atlanta, Georgia
  - Research Site 139, Atlanta, Georgia
  - Research Site 115, Louisville, Kentucky
  - Research Site 129, Detroit, Michigan
  - Research Site 121, Saint Paul, Minnesota
  - Research Site 110, Las Vegas, Nevada
  - Research Site 107, New York, New York
  - Research Site 138, Canton, Ohio
  - Research Site 113, Cincinnati, Ohio
  - Research Site 131, Dayton, Ohio
  - Research Site 123, Charleston, South Carolina
  - Research Site 108, Greenville, South Carolina
  - Research Site 136, Nashville, Tennessee
  - Research Site 135, Austin, Texas
  - Research Site 120, Dallas, Texas
  - Research Site 102, Fairfax, Virginia
  - Research Site 112, Fairfax, Virginia
  - Research Site 105, Spokane, Washington
- Australia (13):
  - Research Site 208, Blacktown, New South Wales
  - Research Site 215, Camperdown, New South Wales
  - Research Site 212, Concord, New South Wales
  - Research Site 217, New Lambton Heights, New South Wales
  - Research Site 201, Sydney, New South Wales
  - Research Site 205, Sydney, New South Wales
  - Research Site 206, Sydney, New South Wales
  - Research Site 216, Waratah, New South Wales
  - Research Site 209, Birtinya, Queensland
  - Research Site 203, Brisbane, Queensland
  - Research Site 210, Gold Coast, Queensland
  - Research Site 202, Nedlands, Western Australia
  - Research Site 207, Nedlands, Western Australia
- China (57):
  - Research Site 319, Hefei, Anhui
  - Research Site 365, Beijing, Beijing Municipality
  - Research Site 310, Beijing, Beijing Municipality
  - Research Site 337, Beijing, Beijing Municipality
  - Research Site 327, Chongqing, Chongqing Municipality
  - Research Site 345, Chongqing, Chongqing Municipality
  - Research Site 353, Chongqing, Chongqing Municipality
  - Research Site 356, Chongqing, Chongqing Municipality
  - Research Site 313, Fuzhou, Fujian
  - Research Site 314, Guangzhou, Guangdong
  - Research Site 322, Guangzhou, Guangdong
  - Research site 367, Guangzhou, Guangdong
  - Research Site 346, Guangzhou, Guangdong
  - Research Site 348, Guangzhou, Guangdong
  - Research Site 350, Guangzhou, Guangdong
  - Research Site 360, Nanning, Guangxi
  - Research Site 334, Baoding, Hebei
  - Research Site 315, Harbin, Heilongjiang
  - Research Site 316, Luoyang, Henan
  - Research Site 317, Xinxiang, Henan
  - Research Site 306, Zhengzhou, Henan
  - Research Site 304, Zhengzhou, Henan
  - Research Site 321, Wuhan, Hubei
  - Research Site 311, Wuhan, Hubei
  - Research Site 309, Changsha, Hunan
  - Research Site 323, Changsha, Hunan
  - Research Site 344, Nanjing, Jiangsu
  - Research Site 305, Nanjing, Jiangsu
  - Research Site 307, Ganzhou, Jiangxi
  - Research Site 349, Nanchang, Jiangxi
  - Research Site 361, Nanchang, Jiangxi
  - Research Site 328, Changchun, Jilin
  - Research Site 301, Changchun, Jilin
  - Research Site 320, Shenyang, Liaoning
  - Research Site 352, Shenyang, Liaoning
  - Research Site 363, Nanjing, Nanjing
  - Research Site 340, Jinan, Shandong
  - Research Site 308, Jinan, Shandong
  - Research Site 333, Linyi, Shandong
  - Research Site 302, Linyi, Shandong
  - Research Site 335, Shanghai, Shanghai Municipality
  - Research Site 326, Shanghai, Shanghai Municipality
  - Research Site 355, Shanghai, Shanghai Municipality
  - Research Site 332, Xi’an, Shanxi
  - Research Site 312, Chengdu, Sichuan
  - Research Site 330, Chengdu, Sichuan
  - Research Site 366, Chengdu, Sichuan
  - Research Site 325, Chengdu, Sichuan
  - Research Site 347, Tianjin, Tianjin Municipality
  - Research Site 318, Tianjin, Tianjin Municipality
  - Research site 368, Tianjin, Tianjin Municipality
  - Research Site 324, Hangzhou, Zhejiang
  - Research Site 329, Hangzhou, Zhejiang
  - Research Site 331, Hangzhou, Zhejiang
  - Research Site 359, Hangzhou, Zhejiang
  - Research site 369, Hangzhou, Zhejiang
  - Research Site 303, Taizhou, Zhejiang
- Taiwan (9):
  - Research Site 408, Kaohsiung City
  - Research Site 405, Kaohsiung City
  - Research Site 406, New Taipei City
  - Research Site 401, Taipei
  - Research Site 402, Taipei
  - Research Site 409, Taipei
  - Research Site 403, Taipei
  - Research Site 407, Taipei
  - Research Site 404, Taoyuan District

IPD SHARING:
Plan to Share IPD: No